CLINICAL TRIAL: NCT04144023
Title: A Phase IB Trial of Neoadjuvant Multi-Epitope HER2 Peptide Vaccine in Patients With HER2-Expressing DCIS
Brief Title: A Vaccine (H2NVAC) Before Surgery for the Treatment of HER2-Expressing Ductal Carcinoma In Situ
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amy C. Degnim, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1713; NCI-2019-07002 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-010561 (Other: Mayo Clinic Institutional Review Board); NCT03793829 (obsolete NCT alias)
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Breast Ductal Carcinoma In Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; Specimen Handling; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (multi-epitope HER2 peptide vaccine H2NVAC, GM-CSF) (Experimental): Prior to standard of care surgery, patients treated at dose levels 1 and 2 receive GM-CSF admixed with multi-epitope HER2 peptide vaccine H2NVAC intradermally on day 1 of each cycle. Treatment repeats every 14 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients treated at dose level 3 receive GM-CSF admixed with multi-epitope HER2 peptide vaccine H2NVAC intradermally on days 1, 4, 8, and 15 for 1 cycle. Patients also undergo ECHO and collection of blood samples throughout the trial and may undergo biopsy on trial.
  Interventions: Biological: Granulocyte-Macrophage Colony-Stimulating Factor; Biological: Multi-epitope HER2 Peptide Vaccine H2NVAC; Procedure: Therapeutic Conventional Surgery; Procedure: Echocardiography Test; Procedure: Biospecimen Collection; Procedure: Biopsy Procedure

INTERVENTIONS:
Biological: Granulocyte-Macrophage Colony-Stimulating Factor — Given intradermally
  Other Names: Colony Stimulating Factor 2; Colony Stimulating Factor, Granulocyte-Macrophage; Colony-Stimulating Factor; Colony-Stimulating Factor 2; CSF; CSF2; GM CSF; GM-CSF; GMCSF; Granulocyte Macrophage Colony Stimulating Factor; Granulocyte Macrophage Colony-Stimulating Factor; Granulocyte-Macrophage Colony Stimulating Factor
Biological: Multi-epitope HER2 Peptide Vaccine H2NVAC — Given intradermally
  Other Names: H2NVAC; HER2 Peptide Vaccine H2NVAC; HER2 Specific Helper T-cell Epitope Vaccine H2NVAC
Procedure: Therapeutic Conventional Surgery — Undergo standard of care surgery
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; ECHOCARDIOGRAPHY; ECHO
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: BIOPSY; BIOPSY_TYPE

SUMMARY:
This phase Ib trial studies the side effects and best dose of a vaccine called H2NVAC before surgery in treating patients with HER2 expressing ductal carcinoma in situ. H2NVAC is a vaccine designed to stimulate specialized white blood cells in hopes of increasing immune response and protecting against breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of multi-epitope HER2 peptide vaccine H2NVAC (H2NVAC) given for 4 treatments in patients with HER2-expressing ductal carcinoma in situ (DCIS) prior to surgery.

II. To determine the dose level of H2NVAC with maximum systemic and intratumoral immunogenicity as measured by activated HER2-specific T lymphocytes or high-affinity antibodies.

SECONDARY OBJECTIVES:

I. To determine intratumoral immunogenicity of H2NVAC in patients with HER2-expressing DCIS.

II. To assess the complete pathological response after 4 treatments of neoadjuvant H2NVAC.

III. To assess the systemic immunogenicity of H2NVAC in patients with HER2-expressing DCIS.

IV. To assess changes in HER2 expression in the DCIS after 4 treatments of neoadjuvant H2NVAC.

V. To assess the distribution of the helper T cell response among T helper cell differentiation states.

OUTLINE: This is a dose-escalation study of multi-epitope HER2 peptide vaccine H2NVAC followed by a dose expansion study for dose level.

Prior to standard of care surgery, patients treated at dose levels 1 and 2 receive granulocyte macrophage-colony-stimulating factor (GM-CSF) admixed with multi-epitope HER2 peptide vaccine H2NVAC intradermally on day 1 of each cycle. Treatment repeats every 14 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients treated at dose level 3 receive GM-CSF admixed with multi-epitope HER2 peptide vaccine H2NVAC intradermally on days 1, 4, 8, and 15 for 1 cycle. Patients also undergo echocardiography (ECHO) and collection of blood samples throughout the trial and may undergo biopsy on trial.

After completion of study treatment, patients are followed up at 3, 6, and 12 months after surgery and optionally at 18 and 24 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must not have received any prior therapy for current DCIS

  * Note: Patients who received tamoxifen, raloxifene, aromatase inhibitor or another agent for prevention of breast cancer may be included as long as the patient has discontinued the treatment at least 2 months prior to baseline study biopsy if they chose to have this collected
  * Note: Concurrent use of endocrine therapy during the vaccination/preoperative period is not allowed. However, standard adjuvant endocrine therapy with tamoxifen or aromatase inhibitor after completion of vaccination and surgery is allowed
* Any degree of HER2 expression as performed on the diagnostic clinical biopsy defined by immunohistochemistry +1, +2, or +3
* Histologically confirmed un-resected operable ductal carcinoma in situ with no evidence of lymph node involvement or distant metastasis

  * Note: suspected microinvasion or definite microinvasion (< 0.1 mm invasion) on core biopsy is allowed
* Patients will be asked to have an additional research biopsy prior to the first vaccination. This is not mandatory for participation
* Patients must have evidence of at least 0.5 cm of disease extent based on mammogram, ultrasound, or magnetic resonance (MRI) imaging
* Absolute neutrophil count (ANC) >= 1500/mm^3 (less than or equal to 28 days prior to registration)
* Platelet count >= 75,000/mm^3 (less than or equal to 28 days prior to registration)
* Hemoglobin >= 9.0 g/dL (less than or equal to 28 days prior to registration)
* Creatinine =< 2 x upper limit of normal (ULN) (less than or equal to 28 days prior to registration)
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2 x ULN (less than or equal to 28 days prior to registration)
* Albumin >= 3 g/dL (less than or equal to 28 days prior to registration)
* Negative serum pregnancy test done =< 7 days prior to Registration, for women of childbearing potential only
* Willing to employ adequate contraception from the time of Registration through 6 months after the final vaccine cycle

  * Note: Adequate contraception methods include birth control pills, barrier device, intrauterine device, or abstinence
* Capable of understanding the investigative nature, potential risks, and benefits of the study
* Capable of providing valid informed consent
* Willing to return to enrolling institution for all study visits (immunizations, blood draws, etc)
* Willing to provide blood samples for correlative research purposes
* Willing to receive a tetanus vaccination if subject has not had one within the past year

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women unwilling to stop breast feeding
  * Women of child bearing potential who are unwilling to employ adequate contraception from the time of registration through 6 months after the final vaccine cycle
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients including patients known to be human immunodeficiency virus (HIV) positive or those on chronic steroids, unless physiologic replacement for adrenal or pituitary insufficiency

  * Note: Must be off systemic steroids greater than or equal to 90 days prior to Registration. However, topical steroids, inhalants or steroid eye drops are permitted
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Uncontrolled acute or chronic medical conditions including, but not limited to the following:

  * Active infection requiring antibiotics
  * Congestive heart failure with New York Heart Association class III or IV moderate to severe objective evidence of cardiovascular disease
  * Myocardial infarction or stroke less than or equal to 6 months prior to registration
* Receiving any other investigational agent
* Other active malignancy at time of registration or less than or equal to the last three years prior to registration. EXCEPTIONS: Non-melanoma skin cancer or carcinoma-in-situ (e.g. of cervix, prostate)

  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment (cytotoxics, monoclonal antibodies, small molecule inhibitors) for their cancer
* Known history of active autoimmune disease that has required systemic treatment in the ≤ 30 days (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) prior to pre-registration

  * NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Patients with vitiligo, Graves' disease, or psoriasis not requiring systemic treatment within the past 30 days are not excluded. Patients with Celiac disease controlled with diet modification are not excluded
* Any prior hypersensitivity or adverse reaction to GM-CSF
* History of trastuzumab-related cardiac toxicity requiring interruption or discontinuation of therapy, even if left ventricular ejection fraction (LVEF) fully recovered
* Baseline LVEF with a value below 55%
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* History of myocardial infarction =< 168 days (6 months) prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life threatening ventricular arrhythmias
* History of ipsilateral radiation to the current affected breast with DCIS

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 2 years
  Number of adverse events reported, measured using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0
Dose limiting toxicities | 14 days post vaccination, 2 years
  Measured using criteria from the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 with grade >= 3 allergic reaction, grade >= 3 autoimmune reaction (except for autoimmune encephalitis grade >=4), grade >= 3 injection site reaction manifesting as an ulceration, grade >= 3 neurologic problem, grade >= 3 non-hematologic or cardiac toxicity, or changes in left ventricular ejection fraction (LVEF) as specified per protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Amy C. Degnim, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials